CLINICAL TRIAL: NCT03961555
Title: A Phase 2b Randomized Blinded Study to Evaluate SYN023 Compared to Human Rabies Immune Globulin in Post Exposure Prophylaxis of Rabies in Adults With Different Rabies Exposure Risks
Brief Title: Comparison of SYN023 to Human Rabies Immune Globulin in Post Exposure Prophylaxis of Rabies
Acronym: ARPEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synermore Biologics Co., Ltd. (Industry)
Collaborators: Synermore Biologics USA Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SYN023-004
Record Dates: First submitted 2019-05-16; First posted 2019-05-23 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2023-05

CONDITIONS: Rabies
Keywords: Post-exposure prophylaxis of Rabies
MeSH Terms: conditions — Rabies | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Risk Group: SYN023+Rabies vaccine (Experimental): The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). Bites to the head, neck, genitalia arm or hand are not included in the LRG. The initial 20 subjects in the LRG were to be randomized on a 3:1 (SYN023 to Human Rabies Immune Globulin (HRIG)) ratio. The general 60 subjects in the LRG were to be allocated with a 1:1 randomization to either SYN023 or HRIG treatment arms.
  SYN023:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 0.3 mg/kg of SYN023
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: Initial LRG subjects received 4 vaccine doses (Days 1, 4, 8,15); General LRG subjects received 5 vaccine doses (Days 1, 4, 8, 15, and 29).
  Interventions: Biological: SYN023; Biological: Rabies vaccine
- Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies vaccine (Active Comparator): The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). Bites to the head, neck, genitalia arm or hand are not included in the LRG. The initial 20 subjects in the LRG were to be randomized on a 3:1 (SYN023 to Human Rabies Immune Globulin (HRIG)) ratio. The general 60 subjects in the LRG were to be allocated with a 1:1 randomization to either SYN023 or HRIG treatment.
  HRIG:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 20 IU/kg
  * Frequency/duration: at Day 1
  Rabies vaccine :
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: Initial LRG subjects received 4 vaccine doses (Days 1, 4, 8,15); General LRG subjects received 5 vaccine doses (Days 1, 4, 8, 15, and 29)
  Interventions: Biological: HRIG (HyperRab); Biological: Rabies vaccine
- Normal Risk Group: SYN023+Rabies vaccine (Experimental): The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). The NRG were consisted of all WHO Category 3 exposure. Subjects were to be allocated with a 1:1 randomization to either SYN023 or Human Rabies Immune Globulin (HRIG) treatment arms.
  SYN023:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 0.3 mg/kg of SYN023
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: at Day 1, 4, 8, 15, 29
  Interventions: Biological: SYN023; Biological: Rabies vaccine
- Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies vaccine (Active Comparator): The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). The NRG were consisted of all WHO Category 3 exposure. Subjects were to be allocated with a 1:1 randomization to either SYN023 or Human Rabies Immune Globulin (HRIG) treatment arms.
  HRIG:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 20 IU/kg
  * Frequency/duration: at Day 1
  Rabies vaccine (RabAvert/Rabipur):
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: at Day 1, 4, 8, 15, 29
  Interventions: Biological: HRIG (HyperRab); Biological: Rabies vaccine

INTERVENTIONS:
Biological: SYN023 — it is administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  Arms: Low Risk Group: SYN023+Rabies vaccine; Normal Risk Group: SYN023+Rabies vaccine
Biological: HRIG (HyperRab) — it is administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  Arms: Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies vaccine; Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies vaccine
Biological: Rabies vaccine — it should be administered in deltoid muscle
  Other Names: RabAvert; Rabipur

SUMMARY:
This is a Phase 2b, double blinded, randomized study of SYN023 compared to HyperRab® (a licensed Rabies immune globulin from human sources, HRIG) for the prevention of rabies as part of post-exposure prophylaxis (PEP). The trial will enroll sequentially two different risk substrata of WHO Category 3 rabies exposure which are Low Risk Group (LRG) and Normal Risk Group (NRG). The enrollment will be stepwise while subject's data will be reviewed by data and safety monitoring board (DSMB) to confirm the safety and permit for next enrollment. Besides, rabies vaccine would be administered within 75 minutes after Study Drug in each group.

This trial is proposed to further the licensure of SYN023 to provide an effective PEP alternative available to those exposed persons who need such a product. A placebo-controlled rabies trial is unethical thus HRIG is selected as the control group. Rabies immune globulin from equine and human sources (HRIG) have been evaluated in many trials and HRIG is the standard of care in the United States.

ELIGIBILITY:
Inclusion Criteria (Low Risk Group):

Subjects must meet all of the following criteria at the time of subject ID assignment:

1. History of dog, cat, mongoose, fox, ferret, skunk, bat or raccoon bite to trunk, leg, ankle or foot, or lick or scratch with, or of broken skin or mucous membrane saliva or neural tissue contamination, unprotected physical bat contact, scratch or saliva contamination of the head or neck without broken skin all ≤ 54 hours
2. Has completed the written informed consent process and signed informed consent document
3. Males and females
4. Is age equal or more than 18 years on Study Day 1
5. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
6. Lives within 2 hour journey by available transportation to study center
7. For female subjects: agrees to avoid pregnancy from Study Day 1 through Study Day 121. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide

Inclusion Criteria (Normal Risk Group)

Subjects must meet all of the following criteria at the time of subject ID assignment:

1. History of dog, cat, mongoose, fox, ferret, skunk, bat or raccoon bite to any body part, lick or scratch with, or of broken skin, mucous membrane saliva or neural tissue contamination, or unprotected physical bat contact all ≤ 54 hours from post exposure prophylaxis (PEP)
2. Has completed the written informed consent process and signed informed consent document.
3. Males and females
4. Is age equal or more than 18 years on Study Day 1
5. Agrees to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and has no current plans to move from the study area for the duration of the study
6. Lives within 2 hour journey by available transportation to study center
7. For female subjects: agrees to avoid pregnancy from agrees to avoid pregnancy from Study Day 1 through Study Day 121. Women physically capable of pregnancy (not sterilized and still menstruating or within 1 year of the last menses if menopausal) in sexual relationships with men must use an acceptable method of avoiding pregnancy during this period. Acceptable methods of avoiding pregnancy include a sterile sexual partner, sexual abstinence (not engaging in sexual intercourse), hormonal contraceptives (oral, injection, transdermal patch, or implant), vaginal ring, intrauterine device (IUD), or the combination of a condom or diaphragm with spermicide

Exclusion Criteria:

Subjects must have had none of the following at the time of subject ID assignment:

1. Clinical evidence of rabies infection
2. Category 3 exposure > 54 hours before Study Drug receipt
3. History or serological evidence of previous rabies vaccination
4. Previous receipt of equine or human rabies globulin
5. History of hypersensitivity reaction to equine or human immunoglobulin.
6. Received immunoglobulin or blood products within 42 days before Study Day 1
7. Received any investigational drug therapy or investigational vaccine within 60 days before Study Day 1
8. Planned participation in any other investigational study during the study period.
9. Receiving systemic immunosuppressant medication such as systemic corticosteroids but not limited to systemic corticosteroids
10. History or laboratory evidence of any past, present, or possible immunodeficiency state including but not limited to any laboratory indication of HIV infection
11. Previous medical history that may compromise the safety of the subject in the study according to the opinion of the principal investigator
12. History or evidence on physical examination of any systemic disease or any acute or chronic illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or activity of SYN023
13. Pregnancy (results of the urine pregnancy test MUST be known before enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Clinical Research Solutions PC -Milan, Milan, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Philippines (9):
  - Baguio General Hospital and Medical Center, Baguio City, Benguet
  - De La Salle Health Sciences Institute Independent Ethics Committee, Cavite City, Calabarzon
  - Southern Philippines Medical Center, Davao City, Davao (Region XI)
  - Manila Doctors Hospital Institutional Review Board, Manila, National Capital Region
  - Asian Hospital and Medical Center, Muntinlupa, National Capital Region
  - Center of Excellence in Drug Research, Evaluation and Studies, Inc., Muntinlupa, National Capital Region
  - Research Institute For Tropical Medicine, Muntinlupa, National Capital Region
  - Far Eastern University Hospital Nicanor Reyes Medical Foundation, Quezon City, National Capital Region
  - Mary Johnston Hospital, Manila

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quiambao BP, Payumo RA, Roa C, Borja-Tabora CF, Emmeline Montellano M, Reyes MRL, Zoleta-De Jesus L, Capeding MR, Solimen DP, Barez MY, Reid C, Chuang A, Tsao E, McClain JB. A phase 2b, Randomized, double blinded comparison of the safety and efficacy of the monoclonal antibody mixture SYN023 and human rabies immune globulin in patients exposed to rabies. Vaccine. 2024 Sep 17;42(22):126018. doi: 10.1016/j.vaccine.2024.05.066. Epub 2024 Jun 4. PMID 38834432

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine: The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). Bites to the head, neck, genitalia arm or hand are not included in the LRG. The initial 20 subjects in the LRG were to be randomized on a 3:1 (SYN023 to Human Rabies Immune Globulin (HRIG)) ratio. The general 60 subjects in the LRG were to be allocated with a 1:1 randomization to either SYN023 or HRIG treatment arms.
  HRIG:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 20 IU/kg
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: Initial LRG subjects received 4 vaccine doses (Days 1, 4, 8,15); General LRG subjects received 5 vaccine doses (Days 1, 4, 8, 15, and 29).
- Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine: The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). The NRG were consisted of all WHO Category 3 exposure. Subjects were to be allocated with a 1:1 randomization to either SYN023 or Human Rabies Immune Globulin (HRIG) treatment arms.
  HRIG:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 20 IU/kg
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: at Day 1, 4, 8, 15, 29
Period: Overall Study
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Started | 45 | 35 | 184 | 184
Completed | 45 | 34 | 178 | 178
Not Completed | 0 | 1 | 6 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 4
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 2 | 2
Not completed — No treatment received | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized by treatment group for all subjects in the As-treated Population. The as-treated population grouped by actual treatment received included all randomly assigned subjects with at least one dose of study treatment.
Groups:
- Low Risk Group: SYN023+Rabies Vaccine: This includes all participants in the Low Risk Group (LRG) receiving SYN023+Rabies Vaccine.
- Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine: This includes all participants in the Low Risk Group (LRG) receiving Human Rabies Immune Globulin (HRIG)+Rabies Vaccine.
- Normal Risk Group: SYN023+Rabies Vaccine: This includes all participants in the Normal Risk Group (NRG) receiving SYN023+Rabies Vaccine.
- Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine: This includes all participants in the Normal Risk Group (NRG) receiving Human Rabies Immune Globulin (HRIG)+Rabies Vaccine.
- Total: Total of all reporting groups
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Total
Number analyzed (Participants) | 45 | 35 | 183 | 184 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (14.26) | 38.4 (13.73) | 31.9 (11.33) | 31.3 (12.49) | 34.9 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 85 | 84 | 211
  Male | 21 | 17 | 98 | 100 | 236
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45 | 35 | 183 | 184 | 447
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 45 | 35 | 183 | 182 | 445
Region of Enrollment [Number; unit: participants]
  Philippines | 45 | 35 | 183 | 184 | 447
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.70 (4.612) | 23.66 (4.732) | 23.89 (4.787) | 23.69 (4.573) | 24.25 (4.664)

OUTCOME MEASURES:

1. Primary Outcome: Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC) at Study Day 8
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Day 8
Population: The primary efficacy analyses were performed and summarized for the for the Normal Risk Group per-protocol population. Results for the Low Risk Group per-protocol population are only presented in-text tables. The per-protocol population included all as-treated subjects without any major protocol deviation who had met all inclusion/exclusion criteria and received complete study treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Number analyzed (Participants) | 40 | 31 | 153 | 156
IU/mL | 4.70 (0.37) | 0.13 (0.10) | 3.30 (0.61) | 0.17 (1.39)

2. Primary Outcome: Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC) at Study Day 99
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Day 99
Population: The primary efficacy analyses were performed and summarized for the for the Normal Risk Group per-protocol population. Results for the Low Risk Group per-protocol population are only presented in-text tables. Per-protocol population: all subjects who were randomly assigned, received the correct study drug, met inclusion/exclusion criteria, completed all rabies scheduled vaccinations, lacked major protocol deviations, had adequate wound treatment and study drug injection of all exposure sites.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Number analyzed (Participants) | 40 | 31 | 153 | 152
IU/mL | 0.66 (1.13) | 1.72 (1.83) | 0.97 (1.21) | 1.47 (1.60)

3. Primary Outcome: Percentage of Participants With Rabies Virus Neutralizing Activity (RVNA) ≥0.5 IU/mL at Study Day 99
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Day 99
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Number analyzed (Participants) | 40 | 31 | 154 | 156
Participants | 30 | 28 | 138 | 142

4. Primary Outcome: Number of Probable or Confirmed Rabies Cases
Description: Case Classification Human Rabies
  * Suspected: A case that is compatible with the clinical case definition
  * Probable: A suspected case (above) plus history of contact with a suspected rabid animal.
  * Confirmed: A suspected case that is laboratory-confirmed.
Time Frame: Day 1 to Day 365
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Number analyzed (Participants) | 40 | 31 | 154 | 156
participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Rabies Virus Neutralizing Activity (RVNA) of Geometric Mean Concentration (GMC) at Study Day 4
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT).
Time Frame: Day 4
Population: The secondary efficacy analyses were performed and summarized for the for the Normal Risk Group per-protocol population. Results for the Low Risk Group per-protocol population are only presented in-text tables. Per-protocol population: all subjects who were randomly assigned, received the correct study drug, met inclusion/exclusion criteria, completed all rabies scheduled vaccinations, lacked major protocol deviations, had adequate wound treatment and study drug injection of all exposure sites.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/mL
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Number analyzed (Participants) | 40 | 30 | 154 | 156
IU/mL | 3.30 (1.27) | 0.12 (0.36) | 3.30 (0.60) | 0.14 (0.82)

6. Secondary Outcome: Area Under the Efficacy Curve for the Geometric Mean Concentration (GMC) of Rabies Virus Neutralizing Activity (RVNA)
Description: Rabies Virus Neutralizing Activity (RVNA) was assessed using Rapid Fluorescent Focus Inhibition Test (RFFIT). Area Under the Efficacy Curve for the GMC of RVNA from Study Day 1 to Day 15 after administration (AUEC1-15)
Time Frame: Day 1 to Day 15
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day.IU/mL
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Low Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: Human Rabies Immune Globulin (HRIG)+Rabies Vaccine
Number analyzed (Participants) | 40 | 31 | 154 | 156
day.IU/mL | 42.91 (0.44) | 5.79 (1.43) | 46.00 (0.57) | 9.81 (2.29)

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The Cmax of CTB011 and CTB012 derived from non-compartmental analysis.
Time Frame: Day 1 to Day 99
Population: The pharmacokinetics of SYN023 was analyzed in the LRG and NRG per-protocol population. No detectable and quantifiable levels of CTB011 and CTB012 were observed in human rabies immune globulin groups, so no PK or statistical analysis was planned.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine
Number analyzed (Participants) | 40 | 154
ng/mL
  Cmax for CTB011 | 903 (23.8) | 700 (25.9)
  Cmax for CTB012 | 916.5 (31.3) | 628 (32.6)

8. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: The Tmax of CTB011 and CTB012 derived from non-compartmental analysis.
Time Frame: Day 1 to Day 99
Population: as for outcome 7
Measure: Median (Full Range); unit: day
Arm/Group | Low Risk Group: SYN023+Rabies Vaccine | Normal Risk Group: SYN023+Rabies Vaccine
Number analyzed (Participants) | 40 | 154
day
  Tmax for CTB011 | 2.93 (0.23) [2.58 to 14.15] | 2.89 (0.34) [2.60 to 13.96]
  Tmax for CTB012 | 2.87 (0.34) [2.58 to 14.02] | 2.89 (0.34) [2.60 to 13.93]

ADVERSE EVENTS:
Time Frame: 365 days
Groups:
- LRG: SYN023+Rabies Vaccine: The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). Bites to the head, neck, genitalia arm or hand are not included in the LRG. The initial 20 subjects in the LRG were to be randomized on a 3:1 (SYN023 to Human Rabies Immune Globulin (HRIG)) ratio. The general 60 subjects in the LRG were to be allocated with a 1:1 randomization to either SYN023 or HRIG treatment arms.
  SYN023:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 0.3 mg/kg of SYN023
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: Initial LRG subjects received 4 vaccine doses (Days 1, 4, 8,15); General LRG subjects received 5 vaccine doses (Days 1, 4, 8, 15, and 29).
- LRG: HRIG+Rabies Vaccine: The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). Bites to the head, neck, genitalia arm or hand are not included in the LRG. The initial 20 subjects in the LRG were to be randomized on a 3:1 (SYN023 to Human Rabies Immune Globulin (HRIG)) ratio. The general 60 subjects in the LRG were to be allocated with a 1:1 randomization to either SYN023 or HRIG treatment arms.
  HRIG:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 20 IU/kg
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: Initial LRG subjects received 4 vaccine doses (Days 1, 4, 8,15); General LRG subjects received 5 vaccine doses (Days 1, 4, 8, 15, and 29).
- NRG: SYN023+Rabies Vaccine: The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). The NRG were consisted of all WHO Category 3 exposure. Subjects were to be allocated with a 1:1 randomization to either SYN023 or Human Rabies Immune Globulin (HRIG) treatment arms.
  SYN023:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 0.3 mg/kg of SYN023
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: at Day 1, 4, 8, 15, 29
- NRG: HRIG+Rabies Vaccine: The subjects were enrolled in the study sequentially into 2 different risk substrata of WHO Category 3 rabies exposure, which included Low Risk Group (LRG) and Normal Risk Group (NRG). The NRG were consisted of all WHO Category 3 exposure. Subjects were to be allocated with a 1:1 randomization to either SYN023 or Human Rabies Immune Globulin (HRIG) treatment arms.
  HRIG:
  * Interventions: are administered by direct injection into the wound or by subcutaneous or intramuscular injection when this is not possible
  * Dosage: 20 IU/kg
  * Frequency/duration: at Day 1
  Rabies vaccine:
  * Interventions: should be administered in deltoid muscle
  * Dosage: 1 mL after reconstitution
  * Frequency/duration: at Day 1, 4, 8, 15, 29
Arm/Group | LRG: SYN023+Rabies Vaccine | LRG: HRIG+Rabies Vaccine | NRG: SYN023+Rabies Vaccine | NRG: HRIG+Rabies Vaccine
All-Cause Mortality (participants affected / at risk) | 0/45 | 1/35 | 0/183 | 0/184
Serious Adverse Events (participants affected / at risk) | 0/45 | 1/35 | 1/183 | 2/184
Other Adverse Events (participants affected / at risk) | 9/45 | 11/35 | 40/183 | 30/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LRG: SYN023+Rabies Vaccine (N=45) | LRG: HRIG+Rabies Vaccine (N=35) | NRG: SYN023+Rabies Vaccine (N=183) | NRG: HRIG+Rabies Vaccine (N=184)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LRG: SYN023+Rabies Vaccine (N=45) | LRG: HRIG+Rabies Vaccine (N=35) | NRG: SYN023+Rabies Vaccine (N=183) | NRG: HRIG+Rabies Vaccine (N=184)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 3
Fatigue (General disorders) | 0 | 0 | 2 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1
Vaccination site pain (General disorders) | 0 | 0 | 0 | 1
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 2 | 4
Urinary tract infection (Infections and infestations) | 2 | 0 | 5 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1
Parasitic gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Viral rash (Infections and infestations) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 3
Eosinophil count increased (Investigations) | 0 | 0 | 6 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Differential white blood cell count abnormal (Investigations) | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 5 | 5
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03961555/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT03961555/SAP_001.pdf